CLINICAL TRIAL: NCT00403910
Title: Phase 3 Study Of Antiremodeling Effect Of Aldosterone Receptors Blockade With Canrenone In Mild Chronic Heart Failure
Brief Title: Antiremodeling Effect Of Aldosterone Receptors Blockade With Canrenone In Mild Chronic Heart Failure. AREA IN-CHF Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heart Care Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 17
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2009-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Canrenone

INTERVENTIONS:
Drug: Canrenone

SUMMARY:
The RALES study has shown that spironolactone reduces the risk of morbidity and mortality both from progressive heart failure and sudden death, in patients with NYHA III or IV heart failure. This favourable effect was clearly independent from a diuretic effect. Antialdosterone drugs may be effective because they opposes the effects of aldosterone on sodium retention, loss of magnesium and potassium, sympathetic activation, baroreceptor function and vascular compliance. Antialdosterone treatment may also antagonize the effect of aldosterone in promoting cardiac fibrosis. In a RALES substudy baseline serum PIIINP, a marker of cardiac fibrosis synthesis showed an independent negative correlation with survival and CHF hospitalizations in the placebo group. Therefore it seems interesting to evaluate the effect of an Aldosterone receptor blocker on progression of left ventricular dysfunction in patients with mild heart failure assuming standard therapy.

DETAILED DESCRIPTION:
The protocol is sponsored by and independent organization and partially supported by Therabel

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of congestive heart failure in NYHA class II
* Left ventricular ejection fraction <= 45% measured within 6 months from enrolment
* Stable standard heart failure therapy (if patients are on beta blocker drugs, treatment must have been started at least three months before enrolment)
* Informed consent (obtained prior of any study procedures)

Exclusion Criteria:

* Age <18 and >80
* Serum creatinine level > 2.5 mg per deciliter
* Serum potassium level > 5.0 mmol per liter
* Valvular heart disease amenable to surgical treatment
* Congenital heart disease
* Unstable angina and/or acute myocardial infarction and/or coronary revascularization procedure within three months before enrolment
* Intravenous therapy with inotropic drugs within three months before enrolment
* History of resuscitated ventricular fibrillation or tachycardia, unless these occurred within 24 hours of an acute myocardial infarction or the subject has an implanted an automatic cardioverter defibrillator
* Chronic active hepatitis or cirrhosis
* Malignant neoplasm or any life threatening non cardiac disease
* History of hypersensitivity to study drug
* Pregnancy or lactating or childbearing age women who are not protected by an accepted method of contraception
* History of drug or alcohol abuse
* Legal incapacity and/or other circumstances rending the patient unable to understand the nature, scope and possible consequences of the study.
* Evidence of uncooperative attitude
* Any condition other than heart failure that does not permit an optimal participation to the trial
* Participation to other RCTs during the last 3 months
* Treatment with: Lithium salts, Potassium sparing diuretics, oral positive inotropic drugs or any investigational drug

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2002-09; Study Completion 2006-07

PRIMARY OUTCOMES:
Changes in echocardiographic left ventricular diastolic volume

SECONDARY OUTCOMES:
Changes in left ventricular systolic volume
Changes in ejection fraction
Changes in NYHA class
cardiac mortality
hospitalization for cardiac causes
combination of cardiac mortality hospitalizations for cardiac causes

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Boccanelli, MD, Study Chair — Ospedale San Giovanni di Roma
Locations (45):
- Italy (45):
  - Presidio GM Lancisi, Ancona
  - Az Ospedaliera Giuseppe Moscati, Avellino
  - Presidio Ospedaliero Moscati, Aversa (CE)
  - Ospedale Monsignor Angelo R di Miccoli, Barletta (BA)
  - Ospedali Riuniti, Bergamo
  - Cardiologia Tiarini Corticella, Bologna
  - Ospedale Generale Provinciale, Bolzano
  - Az Osp G Brotzu - S Michele, Cagliari
  - Az Ospedaliera S Anna e S Sebastiano, Caserta
  - Ospedale San Raffaele G Giglio, Cefalù (PA)
  - Ospedale Civile San Giuseppe, Empoli (FI)
  - Ospedale Santa Maria del Prato, Feltre
  - Ospedale Civile Dario Camberlingo, Francavilla Fontana (BR)
  - Az Osp-Univ San Martino, Genova
  - Ospedale Civile, Ivrea
  - Ospedale Fatebenefratelli, Milan
  - Hepseria Hospital Modena SPA, Modena
  - Ospedale Policlinico, Modena
  - Fondazione Evangelica Betania, Napoli
  - Ospedale V Cervello, Palermo
  - Presidio Ospedaliero di Passirana, Passirana Rho (MI)
  - Ospedale Policlinico S Matteo IRCCS, Pavia
  - Azienda Ospedaliera di Perugia, Perugia
  - Ospedale della val di nievole, Pescia (PT)
  - Azienda CREAS - IFC CNR San Cartaldo, Pisa
  - Ospedale Generale Provinciale Lotti, Pontedera (PT)
  - Ospedale Civile, Ragusa (RG)
  - Ospedale Infermi, Rimini
  - Ospedale San Camillo, Roma
  - Ospedale Sant'Andrea, Roma
  - Ospedale Santo Spirito, Roma
  - Policlinico Luigi di Liegro, Roma
  - Az Osp San Giovanni di Dio e Ruggi d'Aragona, Salerno
  - Ospedale G Fra Cristoforo, San Bonifacio (VR)
  - Ospedale casa Sollievo della Sofferenza, San Giovanni Rotondo (FG)
  - Presidio Ospedaliero di Saronno, Saronno
  - Ospedale San Bartolomeo, Sarzana (GE)
  - Ospedale SS Annunziata, Sassari
  - IRCCS Policlinico Multimedica, Sesto San Giovanni
  - Fondazione S Maugeri Clinica del Lavoro, Telese Terme (BN)
  - Ospedale Cardinale Panico, Tricase (LE)
  - Az Osp-Univ Ospdali Riuniti, Trieste
  - Ospedale San Luca, Vallo Della Lucania (SA)
  - Ospedale di Circolo e Fondazione Macchi, Varese
  - Ospedali Civili Riuniti, Venezia

REFERENCES:
- [Background] Cacciatore G, Boccanelli A, Mureddu GF, Maggioni AP, Latini R, Masson S, de Simone G; Investigatori dell' Area In-CHF. [The AREA IN-CHF trial (antiremodeling effect of aldosterone receptors blockade with canrenone in mild chronic heart failure): rationale and design]. Ital Heart J. 2005 May;6 Suppl 1:66S-74S. Italian. PMID 15945301
- [Background] de Simone G, Chinali M, Mureddu GF, Cacciatore G, Lucci D, Latini R, Masson S, Vanasia M, Maggioni AP, Boccanelli A; AREA-in-CHF Investigators. Effect of canrenone on left ventricular mechanics in patients with mild systolic heart failure and metabolic syndrome: the AREA-in-CHF study. Nutr Metab Cardiovasc Dis. 2011 Oct;21(10):783-91. doi: 10.1016/j.numecd.2010.02.012. Epub 2010 Jun 17. PMID 21939839
- [Background] Clemenza F, Masson S, Conaldi PG, Di Carlo D, Boccanelli A, Mureddu GF, Gonzini L, Lucci D, Maggioni AP, Di Lenarda A, Nicolis EB, Vanasia M, Latini R; AREA IN-CHF Investigators. Galectin-3 and the Mineralocorticoid Receptor Antagonist Canrenone in Mild Heart Failure. Circ J. 2017 Sep 25;81(10):1543-1546. doi: 10.1253/circj.CJ-17-0656. Epub 2017 Aug 31. PMID 28855452
- [Result] Boccanelli A, Mureddu GF, Cacciatore G, Clemenza F, Di Lenarda A, Gavazzi A, Porcu M, Latini R, Lucci D, Maggioni AP, Masson S, Vanasia M, de Simone G; AREA IN-CHF Investigators. Anti-remodelling effect of canrenone in patients with mild chronic heart failure (AREA IN-CHF study): final results. Eur J Heart Fail. 2009 Jan;11(1):68-76. doi: 10.1093/eurjhf/hfn015. PMID 19147459
- [Result] Boccanelli A, Cacciatore G, Mureddu GF, de Simone G, Clemenza F, De Maria R, Di Lenarda A, Gavazzi A, Latini R, Masson S, Porcu M, Vanasia M, Gonzini L, Maggioni AP. Baseline characteristics of patients recruited in the AREA IN-CHF study (Antiremodelling Effect of Aldosterone Receptors Blockade with Canrenone in Mild Chronic Heart Failure). J Cardiovasc Med (Hagerstown). 2007 Sep;8(9):683-91. doi: 10.2459/JCM.0b013e3281053a9a. PMID 17700397